CLINICAL TRIAL: NCT07034781
Title: An Open-label, 2-arm, Single-sequence, Single Oral Dosing, Crossover Clinical Trial to Evaluate Safety and the Pharmacokinetics Between Dapagliflozin, Linagliptin and Metformin in Healthy Adult Subjects
Brief Title: A Study to Evaluate the Safety and Pharmacokinetics of Dapagliflozin, Linagliptin, and Metformin in Healthy Adults
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: AJU Pharm Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 24-IP012
Record Dates: First submitted 2025-06-12; First posted 2025-06-24 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Type2 Diabetes Mellitus
MeSH Terms: interventions — Drug Evaluation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Two-period, single-dose, crossover study
  Interventions: Drug: Comparator 1; Drug: Comparator 2; Drug: Test Drug
- Group B (Experimental): Two-period, single-dose, crossover study (reversed order)
  Interventions: Drug: Comparator 1; Drug: Comparator 2; Drug: Test Drug

INTERVENTIONS:
Drug: Comparator 1 — Dapagliflozin 10mg + Linagliptin 5mg
Drug: Comparator 2 — Metformin 1000mg
Drug: Test Drug — Fixed-dose combination tablet (AJU-A53)

SUMMARY:
To Evaluate the Safety and Pharmacokinetics of Dapagliflozin, Linagliptin, and Metformin in Healthy Adults

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult volunteers aged 19 to 50 years at the time of screening.
* Body mass index (BMI) between 18.0 and 30.0 kg/m², inclusive.

  * Male subjects must weigh ≥50 kg.
  * Female subjects must weigh ≥45 kg.
* No clinically significant congenital or chronic diseases requiring treatment, based on medical history and physical examination.
* Clinically acceptable results from laboratory tests (e.g., hematology, biochemistry, serology, urinalysis) and electrocardiogram (ECG) at screening, as determined by the investigator.
* Willing to use medically accepted contraception (excluding hormonal methods) from the first dose until 50 days after the last dose, and agrees not to donate sperm or eggs during this period.
* Able and willing to provide written informed consent after receiving a full explanation of the study.

Exclusion Criteria:

* Use of drugs known to induce or inhibit drug-metabolizing enzymes within 30 days prior to the first dose, or any medication likely to interfere with the study within 10 days prior to dosing.
* Participation in any clinical trial involving investigational products within 6 months prior to the first dose.
* Whole blood donation within 8 weeks, or component blood donation within 2 weeks prior to the first dose.
* History of gastrointestinal surgery that may affect drug absorption (excluding appendectomy and hernia repair).
* History of excessive alcohol consumption within 1 month prior to the first dose:

  * >21 drinks/week for males, >14 drinks/week for females (1 drink = 50 mL soju, 30 mL whiskey, or 250 mL beer)
* Known hypersensitivity to any component of the investigational product.
* Clinically significant renal, hepatic, cardiovascular, respiratory, metabolic, or infectious diseases, including but not limited to:

  * Moderate to severe renal impairment (eGFR or creatinine clearance <45 mL/min)
  * Dialysis
  * Acute or unstable heart failure
  * Acute myocardial infarction, septicemia, or shock
  * Type 1 diabetes, metabolic acidosis, or history of diabetic ketoacidosis
  * Major surgery planned during the study (except minor procedures not affecting food or fluid intake)
  * Severe infections, trauma, or nutritional deficiencies
* Positive pregnancy test or currently breastfeeding (for female subjects).
* History of significant psychiatric illness.
* Determined by the investigator to be unsuitable for the study for any other reason.

Ages: 19 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Cmax of Dapagliflozin | 0 hour ~ 48 hour after drug administration
  To assess the maximum observed plasma concentration (Cmax) of Dapagliflozin
AUCt of Dapagliflozin | 0 hour ~ 48 hour after drug administration
  To assess the area under the plasma concentration-time curve from time 0 to the last measurable concentration (AUCt) of Dapagliflozin
Cmax of Linagliptin | 0 hour ~ 72 hour after drug administration
  To assess the maximum observed plasma concentration (Cmax) of Linagliptin
AUCt of Linagliptin | 0 hour ~ 72 hour after drug administration
  To assess the area under the plasma concentration-time curve from time 0 to the last measurable concentration (AUCt) of Linagliptin
Cmax of Metformin | 0 hour ~ 48 hour after drug administration
  To assess the maximum observed plasma concentration (Cmax) of Metformin
AUCt of Metformin | 0 hour ~ 48 hour after drug administration
  To assess the area under the plasma concentration-time curve from time 0 to the last measurable concentration (AUCt) of Metformin

CONTACTS AND LOCATIONS:
Locations (1):
- Chung-Ang University Gwangmyeong Hospital, Gwangmyeong, Gyeonggi-do, South Korea